

## STATISTICAL AND EPIDEMIOLOGICAL ANALYSIS PLAN (SEAP) FOR NON-INTERVENTIONAL STUDIES (NIS)


| Document Number: | c38948754-01 |
|---|---|
| BI Study Number: | 1160-0308 |
| BI Investigational Product(s) | Pradaxa |
| Title: | Statistical and Epidemiological Analysis Plan (SEAP) for post-<br>authorization safety study (PASS) to assess the safety and<br>effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese<br>patients with non-valvular atrial fibrillation and concomitant coronary<br>artery disease |
| Brief lay title: | A study based on Japanese medical records that looks at bleeding events in people with atrial fibrillation and coronary artery disease who start taking either dabigatran, rivaroxaban, or warfarin |
| SEAP version identifier: | 1.0 |
| Date of last version of SEAP: | Not applicable |
| NIS Statistician [SEAP author] | |
| NIS [SEAP reviewer] | |
| NIS Data [SEAP reviewer] | |

Proprietary confidential information

© 2022 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 1. TABLE OF CONTENTS

| TITL | LE PAGE | 1 |
|------|---------------------------------------|---|
| 1. | TABLE OF CONTENTS | 2 |
| 2. | LIST OF ABBREVIATIONS | 4 |
| 3. | RESPONSIBLE PARTIES : | 5 |
| 4. | PURPOSE AND SCOPE. | 5 |
| 5. | AMENDMENTS AND UPDATES | 7 |
| 6. | RESEARCH QUESTION AND OBJECTIVE | 7 |
| 7. | RESEARCH METHODS | 3 |
| 7.1 | STUDY DESIGN | 3 |
| 7.2 | SETTING | 3 |
| 7 | 2.1 Follow up period | 3 |
| 7.3 | STUDY POPULATION | |
| 7.4 | STUDY VISITS 10 | ) |
| 8. | VARIABLES | 1 |
| 8.1 | EXPOSURES | |
| 8.2 | | |
| 8 | 2.2.1 Primary outcomes 1 | |
| 8 | Secondary outcomes | 1 |
| | | l |
| 8.3 | COVARIATES | |
| 9. | DATA SOURCES | |
| 10. | DATA MANAGEMENT AND SOFTWARE/TOOLS 13 | |
| 10.1 | | |
| | 2 HANDLING OF MISSING VALUES | |
| 10.3 | | |
| | DATA ANALYSIS | |
| 11.1 | MAIN ANALYSIS | 1 |
| 11.0 | | |
| 11.3 | | |
| 12. | QUALITY CONTROL 10 | |
| 13. | REFERENCES | |
| 13.1 | | |
| 13.2 | 2 UNPUBLISHED REFERENCES | 5 |

# **BOEHRINGER INGELHEIM Group of Companies**Statistical and Enidemiological Analysis Plan (SEAP) for Non

| Statistical and Epidemiological Analysis Flan (SEAF) for Non- | c38948754-01 |
|---|---|
| Interventional Studies (NIS) | |
| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its aff | iliated companies |
| ANNEX 1. LIST OF RECEIPT CODE FOR OAC | 16 |
| ANNEX 2. CODE USED TO CREATE STUDY POPULATION | 17 |
| ANNEX 3. CODE USED FOR OUTCOMES | 21 |
| ANNEX 4. STUDY COVARIATES | 23 |
| ANNEX 5. ANALYSIS TABLE SHELLS | 25 |
| ANNEX 6. REVIEWERS AND APPROVAL SIGNATURES | 32 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

BI Boehringer Ingelheim
CI Confidence Interval
IQR Interquartile range

NIS Non-interventional study

SEAP Statistical and epidemiological analysis plan

DMRP Data management and review plan

AE Adverse Event AF Atrial Fibrillation

ASD Absolute Standardized Difference

CA Competent Authority
CAD Coronary Artery Disease
CCDS Company Core Data Sheet

CHA2DS2- Congestive heart failure, Hypertension, Age ≥ 75 years, Diabetes

VASc mellitus, Stroke, Vascular disease, Age 65-74 years, Sex category (female)

CI Confidence Interval
CML Local Clinical Monitor
CRA Clinical Research Associate

CRF Case Report Form CTP Clinical Trial Protocol

DMRP Data Management and Review Plan
Diagnosis Procedure Combination

eCRF Electronic Case Report Form

ENCePP European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

EMA European Medicines Agency
ESC European Society of Cardiology
FDA Food and Drug Administration

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GI Gastrointestinal

GPP Good Pharmacoepidemiology Practice

GVP Good Pharmacovigilance Practices

HAS-BLED Hypertension, Abnormal renal/liver function, Stroke, Bleeding history or

predisposition, Labile INR, Elderly (>65 years), Drugs/alcohol

concomitantly

HR Hazard Ratio

IB Investigator's Brochure

ICD-10 The 10<sup>th</sup> Revision of the International Classification of Diseases

ICH Intracranial Hemorrhage

ID Identification Number

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

IEC Independent Ethics Committee

IPTW Inverse Probability of Treatment Weighting

IRB Institutional Review Board

MAH Marketing Authorization Holder

MedDRA Medical Dictionary for Regulatory Activities

MI Myocardial Infarction
NIS Non-Interventional Study

NOAC Non-vitamin K Oral Anticoagulant NVAF Non-valvular Atrial Fibrillation

SE Systemic Embolism

VAF Valvular Atrial Fibrillation ESRD End-stage renal disease OAC Oral Anticoagulation

### 3. RESPONSIBLE PARTIES

NIS Statistician [SEAP author]:

SEAP reviewers are:

- BI NIS [SEAP reviewer] (in all cases):
- NIS Data [SEAP reviewer] (in all cases):
- RWE CoE [SEAP reviewer] (for all globally initiated studies and for local studies) involving BI products and Global NIS not involving BI products:
- TM Epi [SEAP reviewer] (When BI NIS is not TM Epi; in all cases):

#### 4. PURPOSE AND SCOPE

SEAP reviewers are expected to be familiar with the NIS protocol entitled "Comparative safety and effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD)" version 1.0 dated 15 November 2021 unless otherwise stated.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
The SEAP addresses the details of the implementation of this study. In the SEAP, you can find
the detailed definitions on how to identify each of the index medication cohorts, detailed data
analysis plan such as the inverse probability of treatment weighting (IPTW), propensity score
matching and main analysis plan.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. AMENDMENTS AND UPDATES

None

### 6. RESEARCH QUESTION AND OBJECTIVE

This non-interventional cohort study using data from large Japan clinical database to access the safety and effectiveness of oral anticoagulants among patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD).

#### **Primary objective:**

To compare the risk of major bleeding between dabigatran and warfarin, and between rivaroxaban and warfarin, among Japanese NVAF patients with concomitant CAD.

#### **Secondary objective:**

To compare the net clinical benefits of dabigatran vs. warfarin, and rivaroxaban vs. warfarin, among Japanese NVAF patients with concomitant CAD. The net clinical benefits are defined as free of composite outcome of stroke/SE/MI/all-cause mortality (inpatient)/major bleeding/major GI bleeding (hospitalization due to GI bleeding)/ICH.

#### **Further objective:**

If the required sample size can be fulfilled and the baseline characteristics are balanced between dabigatran and rivaroxaban groups after IPTW adjustment, to compare the safety and net clinical benefits of dabigatran vs rivaroxaban among Japanese NVAF patients with concomitant CAD.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RESEARCH METHODS

#### 7.1 STUDY DESIGN

This study will be a non-interventional cohort study based on existing data, the ) database. It contains comprehensive medical record data, blood test result data and insurance claims data. Patients meeting the in/exclusion criteria will be selected and will be defined as 3 patient groups:

Group 1: new users of warfarin Group 2: new users of dabigatran Group 3: new users of rivaroxaban

Comparative analyses of the study will follow a two-step approach. In the first step, the primary and secondary outcomes, as well as baseline characteristics, will be compared between Group 1&2 and Group 1&3, respectively.

The second step will utilize the estimated results from step one, which are HRs of major bleeding events between Group 1&2 and between Group 1&3 among NVAF patients with concomitant CAD, to carry out a more accurate sample size calculation to compare dabigatran versus rivaroxaban. If feasible, comparisons will be made on the same outcomes as in step one.

#### 7.2 SETTING

Study Period: the entire time period that includes the look-back period, the cohort entry date (drug index date), and follow-up period for the study population. The study period will be from April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).

Patient Selection Period: the time period for which patients are eligible to enter the cohort, which is from April 18th, 2012 to December 31st, 2020.

Cohort Entry Date: The drug index date, defined as the first date of prescription for dabigatran, rivaroxaban, or warfarin during the patient selection period.

Look-back Period: the 365-day period that ends 1 day prior to the cohort entry date. The earliest start date of the look-back period is April 18th, 2011.

Loss of follow-up: the last data point available in the database during the study period.

#### 7.2.1 Follow up period

The follow up period starts from cohort entry date (first prescription of the drug of interest) and ends at the earliest date of the following dates:

· Discontinuation date of index OAC.

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Discontinuation of the index OAC, defined as a continuous gap of 45 days or more between the expected refill date and the actual refill date. The discontinuation date is defined as 45 days after the expected refill date. The codes for index OAC are listed in Annex 1.

- Date of switching to another OAC.
  - If the index OAC is discontinued, the date of switching to another OAC was the first prescription date of another OAC within 45 days of the expected refill date of the index OAC. The codes of another OAC are the codes in <u>Annex 1</u> excluding codes of the index OAC.
- · Loss of follow-up date.
  - The date of the last inpatient/outpatient encounter during period starting from index OAC date and ending on December 31st, 2020.
- Date of the first occurrence of outcomes of interest (for primary outcome: major bleeding; for secondary outcome: the onset of the first occurring component event; for further outcomes: the respective onset of component events) during period starting from index OAC date and ending on December 31st, 2020.
- Date of death during period starting from index OAC date and ending on December 31st, 2020.
- End of study period date (December 31st, 2020).

#### 7.3 STUDY POPULATION

The target population of the study are Japanese NVAF patients with concomitant CAD, who are prescribed with dabigatran, rivaroxaban, or warfarin. The study population will be selected based on the following in/exclusion criteria:

#### Inclusion Criteria

- 1.  $\geq$ 18 years of age on index date
- 2. Has one year of look-back period prior to the index date (defined as the first date of prescription for dabigatran, rivaroxaban, or warfarin during the study period)
- 3. New users of warfarin, dabigatran, and rivaroxaban, defined as patients without historic use of any oral anticoagulants during the look-back period
- 4. Has at least 1 diagnosis of NVAF during the look-back period prior to or on the index date
- 5. Has at least 1 diagnosis of CAD during the look-back period prior to or on the index date

#### **Exclusion Criteria**

- 1. Diagnosed with end-stage renal disease (ESRD), or undergo hemodialysis, or experience pregnancy during the study period
- 2. Initiate warfarin, dabigatran, rivaroxaban due to valvular AF (VAF), AF associated with mechanical valve malfunction or mechanical complication of heart valve prosthesis, or rheumatic AF
- 3. Underwent joint replacement procedures or diagnosed with venous thromboembolism during the look-back period prior to or on the index date
- 4. Prescribed with more than 1 OAC on the index date

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 5. Prescribed with more than 2 anti-platelet drugs per prescription (triple or quadruple antiplatelet use), or prescribed with any anti-platelet injection
- 6. Patients with missing or ambiguous age or sex information

The codes for OAC are listed in <u>Annex 1</u> and codes to select study population (in/exclusion criteria) are listed in <u>Annex 2</u>.

NVAF during the look-back period prior to or on the index date is defined as patients had diagnosis of AF and had no diagnosis of VAF during the specific period.

Pregnancy during the study period is defined as patients had any of the following:

- · Confirmed diagnosis of pregnancy in the study period.
- In FF1 data (discharge summary data), the admission date was within the study period, and returned true for the pregnancy flag or the number of weeks of pregnancy at the time of hospitalization greater than 0 or the number of weeks of pregnancy at the time of delivery greater than 0.
- · Medical treatment of pregnancy in the study period.

AF associated with mechanical valve malfunction or mechanical complication of heart valve prosthesis is defined as a record with diagnosis of AF and diagnosis of mechanical valve malfunction or mechanical complication of heart valve prosthesis.

Rheumatic AF is defined as a record with diagnosis of AF and diagnosis of rheumatic heart disease.

#### 7.4 STUDY VISITS

Not applicable.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. VARIABLES

Study variables are explained the study protocol section 9.3. you can find operational definitions below:

#### 8.1 EXPOSURES

Respectively for Group 1 (new users of warfarin), group 2 (new users of dabigatran), and group 3 (new users of rivaroxaban), the first prescribed dates of warfarin, dabigatran and rivaroxaban during the study period were selected as the index date, and the patients did not have any OAC prescription during the look back period. The Receipt Code of warfarin, dabigatran and rivaroxaban are in Annex 1.

#### 8.2 OUTCOMES

#### 8.2.1 Primary outcomes

Operational definition of fatal or non-fatal major bleeding is the first new confirmed diagnosis of

blood transfusion (inpatient or outpatient)

OR

- bleeding of inpatient (non-DPC hospital)
- bleeding of inpatient (DPC hospital) with "disease name behind this hospitalization" ("dpcdiseasesegment"=21)

during the follow up period. The ICD-10 diagnosis codes of blood transfusion and bleeding are in Annex 3.

#### 8.2.2 Secondary outcomes

Operational definition of composite outcome of stroke/SE/MI/all-cause mortality (inpatient) /major bleeding/major GI bleeding (hospitalization due to GI bleeding)/ICH is the first new confirmed diagnosis of

- Stroke/SE/MI/ Major bleeding (defined as primary outcome)/ICH OR
- Major GI bleeding (hospitalization due to GI bleeding) OR
- · All-cause mortality (inpatient)

during the follow up period. The ICD-10 diagnosis codes of stroke, SE, MI, major bleeding, ICH, major GI bleeding and death are in Annex 3.

Major GI bleeding (hospitalization due to GI bleeding) is the first new confirmed diagnosis of major GI bleeding in inpatient claims from non-DPC hospital or inpatient claims with "disease name behind this hospitalization" ("dpcdiseasesegment"=21) from DPC hospital.

All-cause mortality (inpatient) is:

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Death of discharge status

OR

- Died within 24 hours of admission in FF1 data (discharge summary data) OR
- · Confirmed diagnosis of death in inpatient claims.



#### 8.3 COVARIATES

Please check section 9.3.3. of the study protocol. List of covariates and operational definitions are added to Annex 4.

The HAS-BLED score is calculated as the total points of the following elements (1 point per element) during the baseline period including the index date.

- · Confirmed diagnosis of hypertension
- Dialysis-dependent kidney disease including confirmed diagnosis of hepatic dysfunction or confirmed diagnosis of renal dysfunction or on hemodialysis treatment OR

Confirmed diagnosis of cirrhosis

OR

Renal transplant

OR

Serum creatinine > 200 m mol/L

OR

ALP > 3x upper limit (1050 IU/L) or ALT > 3x upper limit (132 IU/L) or AST > 3x upper limit (114 IU/L)

OR

Bilirubin > 2x upper limit (2.4 mg/dL)

- Confirmed diagnosis of stroke
- · Confirmed diagnosis of bleeding history
- · Age calculated as of index date > 65 years old
- · Confirmed diagnosis of excessive alcohol use

OR

on treatment of excessive alcohol use

OR

on antiplatelet drugs or non-steroidal anti-inflammatory drug

The CHA2DS2-VASc score is calculated as the total points of the following elements during the baseline period including the index date.

- · Confirmed diagnosis of congestive heart failure (1 point)
- Hypertension (1 point) including confirmed diagnosis of hypertension or on any antihypertensive medications
- Age calculated as of index date  $\geq 75$  years old (2 points)

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Diabetes Mellitus (1 point) including confirmed diagnosis of diabetes mellitus or on any anti-hyperglycemia agents or on any insulin treatment
- · Confirmed diagnosis of stroke (2 points)
- Vascular disease including confirmed diagnoses of MI or peripheral arterial disorder (1 point)
- · Age between 65 and 74 (1 point)
- Female (1 point)

The code used to define the elements of HAS-BLED score and CHA2DS2-VASc score are in Annex 4.

#### 9. DATA SOURCES

Please check section 9.4 of the study protocol.

#### 10. DATA MANAGEMENT AND SOFTWARE/TOOLS

Data is stored using the secured Instant Health Data (IHD) platform (https://www.bhei.com/product). The database is accessed through a user and password system. All study details are addressed either in the protocol, SEAP, or DMRP.

#### 10.1 SOFTWARE/TOOLS

The cohort selection, exposure, outcomes, and covariates derivation will be conducted in IHD platform and the data analysis will be run in BI internal server using SAS software 9.4 (SAS Institute, Inc., Cary, NC) or R Studio 3.5.2.

#### 10.2 HANDLING OF MISSING VALUES

The absence of a code for a condition will be interpreted as an absence of the event. If a study variable is totally missing from a database, it is excluded from the analysis of the pooled data.

If a variable is missing for only some of the patients a missing data category will be added and utilized in the analysis.

#### 10.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

For lab values, distribution of each variable will be assessed. The extreme outliers will be treated as missing values, approaches to handling missing values are described in the previous section.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11. DATA ANALYSIS

Please check section 9.7 of the study protocol

#### 11.1 MAIN ANALYSIS

During the first step of the comparative analysis, the baseline characteristics of the individual NOAC groups will be balanced with the warfarin group to account for potential confounding effects through an inverse probability of treatment weighting (IPTW) method. A multinomial logistic regression model will be used to estimate the generalized propensity score (GPS). The treatment membership (warfarin, dabigatran and rivaroxaban) is the dependent variable and all the covariate variables listed in Annex 4 except for "Anti-platelet drugs" and "The number of anti-platelet drugs per prescription" are independent variables in the multinomial logistic regression model, as the two variables can be fully derived from the variable "Anti-platelet use duration". For each patient, we will obtain the estimated GPS vector with components of the probabilities of receiving each treatment (warfarin, dabigatran and rivaroxaban) through the multinomial logistic regression model.

The stabilized IPTW (s-IPTW) will be used to deal with the inflation of type I error and extremely large weight when using regular IPTW. The s-IPTW is calculated as

$$w_i = \frac{\Pr(T = k)}{\Pr(T = k | X = x_i)}$$

for the *i*th patient, where T is the treatment membership and  $x_i$  is the covariates of this patient. The denominator is the kth component of GPS vector of the *i*th patient who was actually in treatment group k and the numerator is the marginal probability of receiving treatment k[R22-1420].

The GPS distributions (density curves, boxplots) of each treatment will be used to examine GPS overlap between the treatment groups. Patients outside of the common support or overlap area for any component of the GPS vector are removed from the analysis. The area of common support is formed by defining boundaries for each component k, k = 1, 2, 3 of the GPS vector [R22-1419]:

$$\begin{split} & Pr(T=k|x)^{low} \\ & = \max[\min(Pr(T=k|x,T=1)), \min(Pr(T=k|x,T=2)), \min(Pr(T=k|x,T=3))] \\ & Pr(T=k|x)^{high} \\ & = \min[\max(Pr(T=k|x,T=1)), \max(Pr(T=k|x,T=2)), \max(Pr(T=k|x,T=3))] \end{split}$$

The distributions of s-IPTW for each treatment group will be examined, the mean s-IPTW is expected to be close to 1. Weight truncation based on the distributions of s-IPTW will be applied if there are extremely high s-IPTW.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. The baseline demographics, risk factors, and clinical characteristics will be compared between the treatment groups (dabigatran vs warfarin, rivaroxaban vs warfarin, dabigatran vs rivaroxaban) using the absolute standardized difference (ASD) pre- and post- s-IPTW to assess the balance of these confounders. A covariate will be considered well balanced if the ASD is below 0.1.

A Cox proportional hazard regression model with s-IPTW will be used to estimate adjusted hazard ratios (aHRs) of treatments (dabigatran vs warfarin, rivaroxaban vs warfarin) and their 95% CIs on primary, secondary, and further outcomes. The treatment membership is the independent variable in the model. A patient will be censored if discontinuation of the index OAC or switching to another OAC or death or loss to follow-up occurred before outcome event. If substantial covariate imbalance between treatment group is noted assessed by a standardized difference >0.1, then the Cox proportional hazard model will be further adjusted by including covariates that are out of balance in the model. A robust sandwich variance estimation of the treatment effect estimates will be used to account for the fact that the pseudo-population size is inflated or deflated relative to the original population and that weights are estimated [P21-02302].

A sensitivity analysis will be performed by restricting the follow-up period to 3 years for Cox regression models on primary and secondary outcomes.



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.3 SAFETY ANALYSIS

Please check section 9.7.3 of the study protocol

## 12. QUALITY CONTROL

Please check section 9.8 of the study protocol

### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

| R22-1420 | Masahiro Sugihara. Survival analysis using inverse probability of treatment weighted methods based on the generalized propensity score. Pharmaceutical Statistics 2010; 9: 21-34 |
|---|---|
| R22-1419 | Lopez MJ, Gutman R. Estimation of causal effects with multiple treatments: a review and new ideas. Statist. Sci. 2017; 32(3): 432-454 |
| P21-02302 | Rishi J Desai, Jessica M Franklin. Alternative approaches for confounding adjustment in observational studies using weighting based on the propensity score: a primer for practitioners. BMJ 2019; 367:15657 |

#### 13.2 UNPUBLISHED REFERENCES

Not applicable.

## ANNEX 1. LIST OF RECEIPT CODE FOR OAC

| OAC | <b>Receipt Code</b> | Description |
|---|---|---|
| | 610450012 | Warfarin K Tablets 1mg [B01A0] |
| | 610460002 | Arefarin Tablets 1mg [B01A0] |
| | 610462024 | Warfarin Potassium Tablets 0.5mg (HD) [B01A0] |
| | 610462025 | Warfarin Potassium Tablets 2mg (HD) [B01A0] |
| | 610463227 | Warfarin Potassium Tablets 0.5mg [B01A0] |
| | 610463228 | Warfarin Potassium Tablets 2mg [B01A0] |
| | 613330001 | Warfarin Potassium Tablets 1mg [B01A0] |
| Warfarin | 613330002 | Warfarin Potassium Tablets 5mg [B01A0] |
| wariarin | 613330003 | Warfarin Tablets 1mg [B01A0] |
| | 613330004 | Warfarin Tablets 5mg [B01A0] |
| | 620000731 | Warfarin Potassium Tablets 1mg (HD) [B01A0] |
| | 620002332 | Warfarin Tablets 0.5mg [B01A0] |
| | 620002472 | Warlin Tablets 0.5mg [B01A0] |
| | 620002473 | Warlin Tablets 1mg [B01A0] |
| | 620811502 | Warfarin K Tablets 1mg (F) [B01A0] |
| | 620811503 | Warfarin K Tablets 1mg (NISSIN) [B01A0] |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confiden | tial information © 2022 Boehr | inger Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|---|
| | 620811507 | Warfarin K Tablets 1mg (TEVA) [B01A0] |
| | 620811510 | Warfarin K Tablets 1mg (TOWA) [B01A0] |
| | 620811511 | Warfarin K Tablets 1mg (NP) [B01A0] |
| | 621480504 | Warfarin K Tablets 0.5mg (TEVA) [B01A0] |
| | 621480506 | Warfarin K Tablets 0.5mg (TOWA) [B01A0] |
| | 621480507 | Warfarin K Tablets 0.5mg (NP) [B01A0] |
| | 621480604 | Warfarin K Tablets 2mg (NP) [B01A0] |
| | 621938101 | Warfarin K Fine Granules 0.2% (NS) [B01A0] |
| | 621940901 | Warfarin K Fine Granules 0.2% (YD) [B01A0] |
| | 622122601 | Warfarin Granules 0.2% [B01A0] |
| Dabigatran | 622043301 | Prazaxa Capsules 75mg [B01E0] |
| Davigatian | 622043401 | Prazaxa Capsules 110mg [B01E0] |
| | 622068301 | Xarelto Tablets 10mg [B01F0] |
| | 622068401 | Xarelto Tablets 15mg [B01F0] |
| Rivaroxaban | 622449101 | Xarelto Fine Granules Packet 10mg [B01F0] |
| Kivaioxabali | 622449201 | Xarelto Fine Granules Packet 15mg [B01F0] |
| | 622829001 | Xarelto OD Tablets 10mg [B01F0] |
| | 622829101 | Xarelto OD Tablets 15mg [B01F0] |
| Apixaban | 622224901 | Eliquis Tablets 2.5mg [B01F0] |
| | 622225001 | Eliquis Tablets 5mg [B01F0] |
| | 622080901 | Lixiana Tablets 15mg [B01F0] |
| Edoxaban | 622576001 | Lixiana OD Tablets 15mg [B01F0] |
| | 622081001 | Lixiana Tablets 30mg [B01F0] |
| Edoxavan | 622576101 | Lixiana OD Tablets 30mg [B01F0] |
| | 622375201 | Lixiana Tablets 60mg [B01F0] |
| | 622576201 | Lixiana OD Tablets 60mg [B01F0] |

### ANNEX 2. CODE USED TO CREATE STUDY POPULATION

#### DIGNOSIS CODE:

| Indication | ICD-<br>10/<br>disease<br>code | Description |
|---|---|---|
| | I48 | Atrial fibrillation and flutter |
| | I48.0 | Paroxysmal atrial fibrillation |
| AF | I48.1 | Persistent atrial fibrillation |
| | I48.2 | Chronic atrial fibrillation |
| | I48.3 | Typical atrial flutter |
| | I48.4 | Atypical atrial flutter |
| | I48.9 | Atrial fibrillation and atrial flutter, unspecified |
| VAF | 8846941 | valvular atrial fibrillation |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential info | ormation © 2022 Boeh | ringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|---|
| 1 y | 4140014 | coronary artery disease |
| | 8831577 | coronary artery heart disease |
| | I20 | Angina pectoris |
| | I20.0 | Unstable angina |
| | I20.1 | Angina pectoris with documented spasm |
| | I20.8 | Other forms of angina pectoris |
| | I20.9 | Angina pectoris, unspecified |
| | I21 | Acute myocardial infarction |
| | I21.0 | Acute transmural myocardial infarction of anterior wall |
| | I21.1 | Acute transmural myocardial infarction of inferior wall |
| | I21.2 | Acute transmural myocardial infarction of other sites |
| | I21.3 | Acute transmural myocardial infarction of unspecified site |
| | I21.4 | Acute subendocardial myocardial infarction |
| | I21.9 | Acute myocardial infarction, unspecified |
| | I22 | Subsequent myocardial infarction |
| | I22.0 | Subsequent myocardial infarction of anterior wall |
| | I22.1 | Subsequent myocardial infarction of inferior wall |
| | I22.8 | Subsequent myocardial infarction of other sites |
| | I22.9 | Subsequent myocardial infarction of unspecified site |
| | I23 | Certain current complications following acute myocardial infarction |
| CAD | 123.0 | Haemopericardium as current complication following acute myocardial infarction |
| | I23.1 | Atrial septal defect as current complication following acute myocardial infarction |
| | 123.2 | Ventricular septal defect as current complication following acute myocardial infarction |
| | 123.3 | Rupture of cardiac wall without haemopericardium as current complication following acute myocardial infarction |
| | I23.4 | Rupture of chordae tendineae as current complication following acute myocardial infarction |
| | I23.5 | Rupture of papillary muscle as current complication following acute myocardial infarction |
| | 123.6 | Thrombosis of atrium, auricular appendage, and ventricle as current complications following acute myocardial infarction |
| | 123.8 | Other current complications following acute myocardial infarction |
| | I24 | Other acute ischaemic heart diseases |
| | I24.0 | Coronary thrombosis not resulting in myocardial infarction |
| | I24.0 | Dressler syndrome |
| | 124.1 | Other forms of acute ischaemic heart disease |
| 1 | 124.8 | Acute ischaemic heart disease Acute ischaemic heart disease, unspecified |
| | 124.9 | Chronic ischaemic heart disease Chronic ischaemic heart disease |
| | 123 | Chronic ischaenne neart disease |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential inform | nation © 2022 Boo | chringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|---|
| | I25.0 | Atherosclerotic cardiovascular disease, so described |
| | I25.1 | Atherosclerotic heart disease |
| | I25.2 | Old myocardial infarction |
| | I25.3 | Aneurysm of heart |
| | I25.4 | Coronary artery aneurysm and dissection |
| | I25.5 | Ischaemic cardiomyopathy |
| | I25.6 | Silent myocardial ischaemia |
| | I25.8 | Other forms of chronic ischaemic heart disease |
| | I25.9 | Chronic ischaemic heart disease, unspecified |
| | N16.5 | Renal tubulo-interstitial disorders in transplant rejection |
| | N18.5 | Chronic kidney disease, stage 5 |
| | T82.4 | Mechanical complication of vascular dialysis catheter |
| | T86.1 | Kidney transplant failure and rejection |
| | | Unintentional cut, puncture, perforation or haemorrhage during surgical and medical care during kidney dialysis |
| | Y60.2 | or other perfusion Foreign object accidentally left in body during surgical and medical care during kidney dialysis or other |
| | Y61.2 | perfusion |
| ESRD | Y62.2 | Failure of sterile precautions during surgical and medical care during kidney dialysis or other perfusion |
| | Y84.1 | Kidney dialysis as the cause of abnormal reaction of the patient, or of later complication, without mention of misadventure at the time of the procedure |
| | Z49 | Care involving dialysis |
| | Z49.0 | Preparatory care for dialysis |
| | Z49.1 | Extracorporeal dialysis |
| | Z49.2 | Other dialysis |
| | Z49 | Care involving dialysis |
| | Z94.0 | Kidney transplant status |
| | Z99.2 | Dependence on renal dialysis |
| | 277.2 | Complications of cardiac and vascular prosthetic |
| | T82 | devices, implants and grafts |
| | T82.0 | Mechanical complication of heart valve prosthesis |
| | T82.1 | Mechanical complication of cardiac electronic device |
| | 104.1 | Mechanical complication of coronary artery bypass and |
| mechanical valve | T82.2 | valve grafts |
| malfunction or | T82.3 | Mechanical complication of other vascular grafts |
| mechanical | T82.4 | Mechanical complication of vascular dialysis catheter |
| complication of | 102.1 | <u> </u> |
| heart valve | T82.5 | Mechanical complication of other cardiac and vascular devices and implants |
| prosthesis | T82.6 | Infection and inflammatory reaction due to cardiac valve prosthesis |
| | T92.7 | Infection and inflammatory reaction due to other cardiac |
| | T82.7 | and vascular devices, implants and grafts |
| | T92 9 | Other specified complications of cardiac and vascular |
| | T82.8 | prosthetic devices, implants and grafts |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | |
|---|---|---|
| | T82.9 | Unspecified complication of cardiac and vascular prosthetic device, implant and graft |
| | 109 | Other rheumatic heart diseases |
| | 109.0 | Rheumatic myocarditis |
| Rheumatic heart | I09.1 | Rheumatic diseases of endocardium, valve unspecified |
| disease | 109.2 | Chronic rheumatic pericarditis |
| | 109.8 | Other specified rheumatic heart diseases |
| | 109.9 | Rheumatic heart disease, unspecified |
| | I26 | Pulmonary embolism |
| | | Pulmonary embolism with mention of acute cor |
| Venous | I26.0 | pulmonale |
| thromboembolism | | Pulmonary embolism without mention of acute cor |
| | I26.9 | pulmonale |
| | | Phlebitis and thrombophlebitis of other deep vessels of |
| | I80.2 | lower extremities |
| | codes | |
| | presented | |
| Pregnancy | in the | |
| | following | |
| | excel file: | |
| | X | |
| | 1160-0308<br>diagnosis_pregnancy.: | |

## PROCEDURE CODE:

| Procedure | Kubun code | Description |
|---|---|---|
| | C102 | Home self-peritoneal irrigation guidance management fee |
| | C102-2 | Home hemodialysis frequent time guidance management |
| | C155 | Automated peritoneal irrigation equipment add-on fee |
| Hemodialysis | J038-2 | Continuous mild blood filtration |
| Tiemodiarysis | J038-21 | Impaired people add-on fee (continuous mild hemofiltration) |
| | J038-22 | Impaired people add-on fee (continuous mild hemofiltration) |
| | K635-3 | Catheter intraabdominal placement for continuous ambulatory peritoneal dialysis |
| | K082-21 | Artificial joint removal (knee) |
| | K082-22 | Artificial joint removal (foot) |
| | K082-23 | Artificial joint removal (finger) |
| | K082-31 | Artificial joint reimplantation add-on fee (knee) |
| Joint | K082-32 | Artificial joint reimplantation add-on fee (foot) |
| replacement | K082-33 | Artificial joint reimplantation add-on fee (finger) |
| replacement | K082-4 | Total joint replacement of autologous costal bone and cartilage |
| | K082-5 | Total artificial talus replacement |
| | K082-6 | Hip prosthesis sliding surface exchange |
| | K083 | Direct traction using steel codes, and others |
| | K083-2 | Arthrodesis for clubfoot using foot plate and pinch bar |
| Pregnancy | K890 | Tuboplasty (tubo-ovarian transplant, tubal bypass procedure and others) |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | |
|---|---|---|
| | K890-2 | Falloposcopic tuboplasty |
| | K890-3 | Laparoscopic salpingoplasty |
| | K891 | Hysterocervicotomy during delivery (including suture) |
| | K892 | Vaginal breech delivery |
| | K893 | Aspiration delivery |
| | K8941 | Outlet/low forceps delivery |
| | K8942 | Middle forceps delivery |
| | K895 | Perineal/vulvar incision and suturing (during delivery) |
| | K8961 | Perineal/vaginal tear suturing (during delivery) (with involvement of the muscular layer) |
| | K8962 | Perineal/vaginal tear suturing (during delivery) (with involvement of the anal) |
| | K8963 | Perineal/vaginal tear suturing (during delivery) (up to vaginal fornix) |
| | K8964 | Suturing of perineal/vaginal tear (associated with rectal tear) (during delivery) |
| | K897 | Endocervical tear suturing (during delivery) |
| | K8981 | Caesarean delivery (emergency cesarean section) |
| | K8982 | Cesarean section (selective cesarean section) |
| | K8983 | Complication add-on fee (hysterotomy) |

### MEDICATION CODE:

| Medication | Receipt Code | Description |
|---|---|---|
| | 620004669 | Shiphnos I.V.Injection 10mg 0.5%2mL [C01D0] |
| | 620008786 | Agilease I.V.Injection 10mg 0.5%2mL [C01D0] |
| | 620008891 | Tohmol I.V.Injection 10mg 0.5%2mL [C01D0] |
| | 620008931 | Persantin I.V.Injection 10mg 0.5%2mL [C01D0] |
| Anti-platelet injection | 620330301 | Dipyridamole I.V.Injection 10mg (ISEI) 0.5%2mL [C01D0] |
| injection | 620330502 | Dipyridamole I.V.Injection 10mg (NICHIIKO) 0.5%2mL [C01D0] |
| | 642170001 | Agilease Injection 0.5%2mL [C01D0] |
| | 642170008 | Tohmol Injection 0.5%2mL [C01D0] |
| | 642170009 | Persantin Injection 0.5%2mL [C01D0] |
| Anti-platelet Drug | codes presented in the following excel file: 1160-0308 Anti-platelet drug.xlsx | |

### **ANNEX 3. CODE USED FOR OUTCOMES**

| Indication ICD-10 code | Description |
|------------------------|-------------|
|------------------------|-------------|

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Blood transfusion | K92.0 | er Ingelheim International GmbH or one or more of its affiliated companies Haematemesis |
|---|---|---|
| 21004 (141101401011 | D50 | Iron deficiency anaemia |
| | 250 | Iron deficiency anaemia secondary to blood loss |
| | D50.0 | (chronic) |
| | D50.1 | Sideropenic dysphagia |
| | D50.8 | Other iron deficiency anaemias |
| | D50.9 | Iron deficiency anaemia, unspecified |
| | D62 | Acute posthaemorrhagic anaemia |
| | D64.9 | Anaemia, unspecified |
| | H35.6 | Retinal haemorrhage |
| | I31.2 | Haemopericardium, not elsewhere classified |
| | I60 | Subarachnoid haemorrhage |
| | | Subarachnoid haemorrhage from carotid siphon and |
| | I60.0 | bifurcation |
| | I60.1 | Subarachnoid haemorrhage from middle cerebral artery |
| | | Subarachnoid haemorrhage from anterior communicating |
| | I60.2 | artery |
| | | Subarachnoid haemorrhage from posterior |
| | I60.3 | communicating artery |
| | I60.4 | Subarachnoid haemorrhage from basilar artery |
| | I60.5 | Subarachnoid haemorrhage from vertebral artery |
| | 160.6 | Subarachnoid haemorrhage from other intracranial |
| | I60.6 | arteries Subarachnoid haemorrhage from intracranial artery, |
| Bleeding | 160.7 | unspecified |
| | 160.8 | Other subarachnoid haemorrhage |
| | 160.9 | Subarachnoid haemorrhage, unspecified |
| | I61 | Intracerebral haemorrhage |
| | I61.0 | Intracerebral haemorrhage in hemisphere, subcortical |
| | I61.1 | Intracerebral haemorrhage in hemisphere, cortical |
| | I61.2 | Intracerebral haemorrhage in hemisphere, unspecified |
| | I61.3 | Intracerebral haemorrhage in brain stem |
| | I61.4 | Intracerebral haemorrhage in cerebellum |
| | I61.5 | Intracerebral haemorrhage, intraventricular |
| | I61.6 | Intracerebral haemorrhage, multiple localized |
| | I61.8 | Other intracerebral haemorrhage |
| | I61.9 | Intracerebral haemorrhage, unspecified |
| | K92.2 | Gastrointestinal haemorrhage, unspecified |
| | M25.0 | Haemarthrosis |
| | M25.00 | Haemarthrosis, multiple sites |
| | M25.01 | Haemarthrosis, shoulder region |
| | M25.02 | Haemarthrosis, upper arm |
| | M25.03 | Haemarthrosis, forearm |
| | M25.04 | Haemarthrosis, hand |
| | M25.05 | Haemarthrosis, pelvic region and thigh |
| | M25.06 | Haemarthrosis, lower leg |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential information | © 2022 Boehringer I | ngelheim International GmbH or one or more of its affiliated companies |
|---|---|---|
| | M25.07 | Haemarthrosis, ankle and foot |
| | M25.08 | Haemarthrosis, other |
| | M25.09 | Haemarthrosis, site unspecified |
| | N92.0 | Excessive and frequent menstruation with regular cycle |
| | R04 | Haemorrhage from respiratory passages |
| | R04.0 | Epistaxis |
| | R04.1 | Haemorrhage from throat |
| | R04.2 | Haemoptysis |
| | R04.8 | Haemorrhage from other sites in respiratory passages |
| | R04.9 | Haemorrhage from respiratory passages, unspecified |
| | R31 | Unspecified haematuria |
| | R58 | Haemorrhage, not elsewhere classified |
| Stroke/SE/MI/ICH/Maj<br>or GI bleeding/Death | codes presented in the following excel file: 1160-0308 stroke_SE_MI_GI_ICH_ | |

## **ANNEX 4. STUDY COVARIATES**

| N | Category | Variables | Definition |
|---|---|---|---|
| 1 | Demographic characteristics | Age | - By year (calculated on index date) |
| | | Gender | - Male, Female |
| 2 | Ischemic and hematologic characteristics | CHA2DS2-VASc score | Codes used to define elements of CHA2DS2-VASc score in the following excel file: 11600308 CHA2DS2_VASc.xlsx |
| | | HAS-BLED score | Codes used to define elements of HAS- BLED score in the following excel file: 1160-0308 HASBLED.xlsx |
| 3 | Comorbidities | Heart failure | ICD-10 diagnosis codes presented |
| | | Peripheral arterial disorder | in the following excel file: |
| | | Hypertension | |
| | | Diabetes | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Propriet | ary confidential information | © 2022 Boehringer Ingelheim International G | mbH or one or more of its affiliated companies |
|---|---|---|---|
| | | Prior stroke/transient | X |
| | | ischemic attack (TIA)/SE | 1160-0308 |
| | | Cerebrovascular disease | Comorbidities.xlsx |
| | | Myocardial infarction | |
| | | Acute Coronary Syndrome | |
| | | Unstable angina | |
| | | Bleeding history | |
| | | Renal dysfunction | |
| | | Hepatic dysfunction | |
| | | Cancers | |
| | | Peptic ulcer disease | |
| | | Obesity | |
| 4 | Co-medications | Anti-platelet drugs | Anti-platelet drugs include aspirin, |
| | | The number of anti-platelet | clopidogrel, ticagrelor and |
| | | drugs per prescription | prasugrel. The number of anti- |
| | | Anti-platelet use duration | platelet drugs is the number of anti-<br>platelet drugs prescribed on the |
| | | Nonsteroidal anti- | earliest prescription date before or |
| | | inflammatory drugs | on the index date during the look |
| | | Gastric secretion inhibitors | back period. Anti-platelet use |
| | | Statins | duration is based on the number of days from the earliest anti-platelet |
| | | Heparins | prescription date to the index date. |
| | | Proton pump inhibitor | Receipt codes presented in |
| | | Antihypertensive drugs | the following excel file: |
| | | | 1160-0308<br>Comedication.xlsx |
| 5 | Medical | Cardioversion procedures | Receipt codes presented in |
| | procedures | Ablation procedures | the following excel file: |
| | | Percutaneous Coronary | ×≡ |
| | | Intervention or Coronary | 1160-0308 Medical |
| | | Artery Bypass Grafting | procedure.xlsx |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ANNEX 5. ANALYSIS TABLE SHELLS**

Note: Table 1, Table 2a, and Table 3 are shown here to exemplify; please find the complete table shells in the attached excel file below



## **Table 1. Patient Flow Diagram**

| | Dabigatran | Rivaroxaban | Warfarin |
|---|---|---|---|
| Total number of patients database 2008-04-01 - 2020-12-31 | | | |
| Patients prescribed with index drug in selection period | | | |
| Patients older than 18 years old at drug index date | | | |
| Have at least 1y look-back prior drug index date | | | |
| New user of Dabigatran or Rivaroxaban or<br>Warfarin, i.e, patients without historic use of<br>any oral anticoagulants during the look-back<br>period | | | |
| Have at least 1 diagnosis of NVAF during the look-back period prior to or on the index date | | | |
| Have at least 1 diagnosis of CAD during the look-back period prior to or on the index date | | | |
| Excluded because of Diagnosis of end-stage renal disease, or undergo hemodialysis, or experience pregnancy during the study period | | | |
| Excluded because of Initiation of warfarin, dabigatran, rivaroxaban due to valvular AF, AF associated with mechanical valve malfunction or mechanical complication of heart valve prosthesis, or rheumatic AF | | | |

## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential information © 2022 Boehringer Ingelheim Inter- | national GmbH or one | or more of its affiliated | companies |
|---|---|---|---|
| Excluded because Underwent joint replacement procedures or diagnosed with venous thromboembolism during the lookback period prior to or on the index date | | | |
| Excluded because of Prescription with more than 1 OAC on the index date | | | |
| Excluded because of Triple or Quadruple Antiplatelet Use or Antiplatelet Injection | | | |
| Excluded because Patients with missing or ambiguous age or sex information | | | |
| Final cohort | | - | |

Table 2a. Baseline Characteristics Comparisons – Dabigatran vs. Warfarin

| | Crude | | | s-IPTW | s-IPTWAdjusted | | | PS-matched | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Da<br>big<br>atr<br>an | Warfari<br>n | Abs.<br>Std.<br>Dif | Dabigatra<br>n | Wa<br>rfar<br>in | Abs.St<br>d.Dif | Dabig<br>atran | Warf<br>arin | Abs.S<br>td.Dif |
| Age | | | | | | | | | |
| mean (sd) | | | | | | | | | |
| median<br>[IQR] | | | | | | | | | |
| ···Min-Max | | | | | | | | | |
| Gender | | | | | | | | | |
| 1 - Male; n<br>(%) | | | | | | | | | |
| 2 - Female;<br>n (%) | | | | | | | | | |
| CHA2DS2-<br>VASc score | | | | | | | | | |
| mean (sd) | | | | | | | | | |
| median<br>[IQR] | | | | | | | | | |
| ···Min-Max | | | | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential | informat | ion © 2022 Boo | ehringer Ing | gelheim Internationa | ıl GmbH | or one or mo | e of its affilia | ated compar | nies |
|---|---|---|---|---|---|---|---|---|---|
| HAS-BLED score | | | | | | | | | |
| ···mean(sd) | | | | | | | | | |
| ···median[IQR<br>] | | | | | | | | | |
| ···Min-Max | | | | | | | | | |
| Heart failure;<br>n (%) | | | | | | | | | |
| Peripheral<br>arterial<br>disorder; n<br>(%) | | | | | | | | | |
| Hypertension;<br>n (%) | | | | | | | | | |
| Diabetes; n<br>(%) | | | | | | | | | |
| Prior<br>stroke/transie<br>nt ischemic<br>attack<br>(TIA)/SE; n<br>(%) | | | | | | | | | |
| Myocardial infarction; n (%) | | | | | | | | | |
| Acute<br>Coronary<br>Syndrome; n<br>(%) | | | | | | | | | |
| Unstable angina; n (%) | | | | | | | | | |
| Bleeding<br>history; n (%) | | | | | | | | | |
| Renal<br>dysfunction; n<br>(%) | | | | | | | | | |
| Hepatic<br>dysfunction; n<br>(%) | | | | | | | | | |
| Cancers; n (%) | | | | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential | informat | ion © 2022 Boo | ehringer Ing | gelheim Internationa | l GmbH | or one or mo | re of its affilia | ated compar | nies |
|---|---|---|---|---|---|---|---|---|---|
| Peptic ulcer<br>disease; n (%) | | | | | | | | | |
| Cerebrovascul<br>ar disease; n<br>(%) | | | | | | | | | |
| Obesity; n (%) | | | | | | | | | |
| Anti-platelet<br>drugs<br>(include<br>aspirin,<br>clopidogrel,<br>ticagrelor,<br>prasugrel); n<br>(%) | | | | | | | | | |
| The number of anti-platelet drugs per prescription (single antiplatelet, dual antiplatelet, none); n (%) | | | | | | | | | |
| single<br>antiplatelet; | | | | | | | | | |
| dual<br>antiplatelet; | | | | | | | | | |
| none; | | | | | | | | | |
| Antiplatelet use duration; n (%) | | | | | | | | | |
| Single Antiplatelet Use: 6 months to 1 year | | | | | | | | | |
| Single<br>Antiplatelet | | | | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential | informat | ion © 2022 Boo | ehringer Ing | gelheim Internationa | l GmbH | or one or mor | e of its affilia | ated compar | nies |
|---|---|---|---|---|---|---|---|---|---|
| Use: 1 month | | | | | | | | | |
| to 6 months | | | | | | | | | |
| Single Antiplatelet Use: <1 month | | | | | | | | | |
| Dual<br>Antiplatelet<br>Use: 6<br>months to 1<br>year | | | | | | | | | |
| Dual Antiplatelet Use: 1 month to 6 months | | | | | | | | | |
| Dual<br>Antiplatelet<br>Use: <1<br>month | | | | | | | | | |
| None | | | | | | | | | |
| Nonsteroidal<br>anti-<br>inflammator<br>y drugs; n (%) | | | | | | | | | |
| Gastric<br>secretion<br>inhibitors; n<br>(%) | | | | | | | | | |
| Statins; n (%) | | | | | | | | | |
| Heparins; n<br>(%) | | | | | | | | | |
| Proton<br>pump<br>inhibitor; n<br>(%) | | | | | | | | | |
| Antihyperten<br>sive drugs; n<br>(%) | | | | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential | informat | 10n © 2022 Boe | ehringer Ing | gelheim Internationa | I GmbH | or one or mor | e of its affilia | ated compan | ies |
|---|---|---|---|---|---|---|---|---|---|
| Cardioversio | | | | | | | | | |
| n | | | | | | | | | |
| procedures; | | | | | | | | | |
| n (%) | | | | | | | | | |
| Ablation | | | | | | | | | |
| procedures; | | | | | | | | | |
| n (%) | | | | | | | | | |
| Percutaneou | | | | | | | | | |
| s Coronary | | | | | | | | | |
| Intervention | | | | | | | | | |
| or Coronary | | | | | | | | | |
| Artery | | | | | | | | | |
| Bypass | | | | | | | | | |
| Grafting; n | | | | | | | | | |
| (%) | | | | | | | | | |

Table 3. Rates and Risks of Fatal/Non-fatal Major Bleeding

| | Comparison 1 | | Comparison 2 | | Comparison 3* | |
|---|---|---|---|---|---|---|
| | Dabig<br>atran | Warfa<br>rin | Rivaro<br>xaban | Warfa<br>rin | Dabig<br>atran | Rivaroxab<br>an |
| Rate | | | | | | |
| Crude | | | | | | |
| Number of patients | | | | | | |
| Number of events | | | | | | |
| Number of person-years | | | | | | |
| Incidence Rate per 1,000 person-years (95% CI) | | | | | | |
| Incidence Proportion (n (%)) | | | | | | |
| s-IPTW adjusted | | | | | | |
| Number of patients | | | | | | |
| Number of events | | | | | | |
| Number of person-years | | | | | | |
| Incidence Rate per 1,000 person-years (95% CI) | | | | | | |
| Incidence Proportion (n (%)) | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

| Proprietary confidential information © 2022 Boehringe | r Ingelheim I | nternational ( | GmbH or one | or more of its | affiliated con | mpanies |
|---|---|---|---|---|---|---|
| PS-matched | | | | | | |
| Number of patients | | | | | | |
| Number of events | | | | | | |
| Number of person-years | | | | | | |
| Incidence Rate per 1,000 person-years (95% CI) | | | | | | |
| Incidence Proportion (n (%)) | | | | | | |
| Hazard ratios | | | | | | |
| s-IPTWAdjusted Hazard Ratio (95% CI, p value) | | | | | | |
| PS Matched Hazard Ratio (95% CI, p value) | | | | | | |

\*Note: comparison 3 will be conducted if sample size is sufficient (see section 9.5 of protocol)

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c38948754-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 6. REVIEWERS AND APPROVAL SIGNATURES

The NIS SEAP must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI<br>product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi* | X | X | X |
| NIS Data Manager | X | X | X |
| RWE CoE | X | X | |

<sup>\*</sup> When BI NIS lead is not TM Epi

**Study Title:** Comparative safety and effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD)

**Study Number: 1160.0308** 

Protocol Version: V1.0

I herewith certify that I agree to the content of the study SEAP and to all documents referenced in the study SEAP.

| Position: | Name/Date: | Signature: |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |